CLINICAL TRIAL: NCT00851968
Title: A Prospective Randomized Controlled Trial of Complete Versus Selective HepaticVascular Clamping in Hepatectomy
Brief Title: A Trial of Complete Versus Selective HepaticVascular Clamping in Hepatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, ShenFeng, vice president of the Eastern Hepatobiliary Surgery Hospotal, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EHBH-RCT-2008-008
Record Dates: First submitted 2009-02-24; First posted 2009-02-26 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatectomy; Selective HepaticVascular Clamping
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pringle's Maneuver (Active Comparator): Patients with HCC received Pringle's Maneuver in hepatectomy.
  Interventions: Procedure: Pringle's Maneuver
- Hemihepatic vascular Clamping (Experimental): Patients with HCC received Hemihepatic vascular Clamping in hepatectomy
  Interventions: Procedure: Hemihepatic vascular Clamping
- portal vein occlusion (Experimental): Patients with HCC received portal vein occlusion in hepatectomy
  Interventions: Procedure: Portal vein occlusion

INTERVENTIONS:
Procedure: Pringle's Maneuver — The entire hilar pedicle was encircled with a rubber tape to perform a Pringle maneuver with a tourniquet.
  Other Names: Pringle's Maneuver group
  Arms: Pringle's Maneuver
Procedure: Hemihepatic vascular Clamping — The portal vein,hepatic artery ,and biliary duct were dissected in the hilum by opening the peritoneal fascia. Either the right or left portal pedicle was isolated and encircled with a tourniquet or clamped with Shatinsky clamp. Separate clamping of accessory left hepatic artery was performed when present in controlling the left hemihepatic portal traid.
  Other Names: Hemihepatic vascular Clamping group
  Arms: Hemihepatic vascular Clamping
Procedure: Portal vein occlusion — The proper hepatic artery was dissected first from the duodenohepatic ligament, portal pedicle was blocked with a rubber encircled through the posterior wall of proper hepatic artery and the bottom of duodenohepatic ligament.When aberrant hepatic arteries emerging from the superior mesenteric artery are found in duodenohepatic ligament ,they should be dissected and kept unobstructed.
  Other Names: Portal vein occlusion group
  Arms: portal vein occlusion

SUMMARY:
Intraoperative bleeding remains a major concern during liver resection. Pringle maneuver is the most frequently used method to occlude inflow blood of the liver.However, experimental and clinical studies have shown than even short periods of clamping produce some degree of ischemia-reperfusion injury that can result in hepatocellular damage,this damage being especially important in patients with abnormal liver parenchyma such as steatosis and cirrhosis. The aim of this study was to evaluate whether the use of selective vascular clamping should be generalized to HCC patients and help to reduce the ischemia-reperfusion injury.

DETAILED DESCRIPTION:
From recent animal studies, it can be easily concluded that I/R injury of the liver may be a significant factor, which can promote the primary liver tumor recurrence and metastasis. If it is a truth in human, there must be a big challenge to the Pringle maneuver which was adopted routinely in hepatectomy in the past years. Pringle maneuver during hepatic resection may do harm to the liver function, make the tumor cell more aggressive and tend to recurrence. It is suggested that further strategies may be needed for the prevention and treatment of I/R injury ,early and late recurrences.Selective hepatic vascular clamping (SVC)such as hemihepatic vascular occlusion have been used to minimize ischemic injury during liver surgery, especially in patients with abnormal liver parenchyma. However,these procedure used is likely to depend on the surgeon's training or preference rather than on objective data, there is not any further reported data or RCT studies conducted about the postoperative outcome ,especially liver function.To address these issues,we designed a prospective randomized controlled trial comparing the complete hepatic vascular clamping (Pringle maneuver) and selective hepatic vascular clamping ( portal vein or hemi-hepatic occlusion) in patients undergoing hepatectomy. The main objective was to compare the liver I/R injury of two procedures to the postoperative liver function. The secondary objective was to evaluate the feasibility, safety, efficacy, amount of hemorrhage,postoperative complications ,disease-free and overall survival rate of the 2 procedures.

ELIGIBILITY:
Inclusion Criteria:

1. with a clinical diagnosis of primary liver cancer, without any adjuvant therapy;
2. age:18-70years;
3. suitable for partial hepatectomy without other malignancies;
4. compensated cirrhosis with Child-Pugh class A, or B.

Exclusion criteria:

1. reject to attend；
2. with any preoperative adjuvant therapy.
3. with intrahepatic or extrahepatic malignancies;
4. cirrhosis with Child-Pugh class C

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
overall survival | 2010

SECONDARY OUTCOMES:
serum alanine aminotransferase (ALT), bilirubin, prothrombin time, serum albumin and pre-albumin on postoperative 1, 3, 7 day, resection rate, procedure-related complications and hospital mortality,expression of HIF and P-, E-, and L-selectin | 2010

CONTACTS AND LOCATIONS:
Overall Officials: Shen feng, MD, Study Chair — Eastern Hepatobiliary Surgery Hospital Affiliated to Second Military Medical University
Locations (1):
- Eastern Hepatobiliary Surgery Hospital, Shanghai, Shanghai Municipality, China